CLINICAL TRIAL: NCT03886064
Title: Scaling-up Packages of Interventions for Cardiovascular Disease Prevention in Selected Sites in Europe and Sub-Saharan Africa. SPICES Study Implementation Phase
Brief Title: Cardiovascular Disease Prevention in Europe and Sub-Saharan Africa
Acronym: Spices_phase_2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: ERCR SPURBO (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 29BRC18.0256_Spices_phase_2
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Cardiovascular Risk Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Only measurement of clinical endpoints at time zero, then at 6, 12, 18 and 24 months and minimal counseling.
- Interventional group (Other): Measurement of clinical endpoints at time zero, then at 6, 12, 18 and 24 months and minimal counseling followed by multi-behavioral intervention adapted to local resources.
  Interventions: Other: Multi-behavioral intervention

INTERVENTIONS:
Other: Multi-behavioral intervention — The interventional group will then meet regularly under the aegis of the trainer to work on modifying each person's risk factors. The one-hour sessions will be scheduled every two weeks for two months and then every month for two months and then every three months until the end of the study (13 sessions). These sessions will be behavior change sessions, focused on goal setting, action planning, and problem solving. Trainers will facilitate these sessions and use motivational interviewing techniques
  Arms: Interventional group

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death in the world. 17.5 million people died in 2012 due to CVD (31% of all causes of death). In Europe more than 50% of deaths are due to CVD. The CVD mortality rate is higher in the lower socio-economic levels. Three quarters of CVD deaths occur in developing countries (LDCs). According to estimates in 2030, CVD will be responsible for more deaths than the sum of infectious, nutritional, maternal and perinatal diseases in developing countries. The lack of an adequate primary care network in developing countries limits the screening and treatment of people with CVRF. As a result, these people do not benefit from appropriate prevention, are diagnosed late and remain disabled or die at a young age, resulting in significant additional costs for families but also at the macroeconomic level.

Cardiovascular risk factor prevention measures (CVRF) have been shown to be effective. Interventions are possible on a large scale (policies against smoking and unfavorable eating habits, promoting physical activity, etc.). Actions are possible at the individual level, both in primary prevention (fight against the FDRCV) and secondary, where many treatments have proven their effectiveness. These interventions are effective and profitable from a macroeconomic point of view. It has been estimated that the cost for such interventions would not exceed 4% of health expenditure in developing countries and 1-2% in rich countries.

The World Health Organization (WHO) stresses the importance of the triad composed by the patient and his family, the community and health professionals. Results are possible only when these three components work together for the same purpose. Many studies show the benefit of people's involvement in care in rich and developing countries.

SPICES project builds on progress in HIV / AIDS treatment in sub-Saharan Africa (SSA) and chronic disease management through the Innovative Care for Chronic Conditions (ICCC Framework), WHO plan. With regard to HIV treatment, these interventions have proven to be effective and cost-effective in many SSA countries, both in terms of disease control and adherence. These data on communicable and infectious diseases seem to be transferable to non-communicable diseases.

These projects were born from the observation that the model of care of the rich countries (individual approach of the patient, centered on the hospital and the specialist with a regular clinical and paraclinical follow-up) could not be transposed to the developing countries, because the limitation of human, technical and financial resources. But also that this model was becoming more and more difficult to maintain in developed countries or resources become limited. New approaches need to be developed to increase the effectiveness of health systems.

A paradigm shift is needed to improve the control of CVD with greater cost-effectiveness.

The SPICES project incorporates the most up-to-date knowledge to improve the prevention and control of CVD in high-, middle- and low-income countries.

Rich countries and developing countries are therefore involved in the study. The selected sites are France, United Kingdom, Belgium, South Africa and Uganda.

Some main axes of the ICCC Framework will be developed in SPICES:

* improve the efficiency of health professionals through the delegation of skills and appropriate training,
* center care around the patient and his family and more generally his caregivers,
* simplify the monitoring and treatment protocols,
* support patients in their community and emphasize prevention, information and patient education.

A first step of observation in the various countries made it possible to make an inventory of fixtures and to target the most adapted interventions.

The following steps are the implementation of these interventions (delegation of skills, information campaign and screening, improve the availability of treatments, measure of strengthening of compliance, etc. ..) and their evaluation.

This study, carried out in France and integrated into the SPICES project, will test the best non-pharmacological interventions selected in the community and by the community.

ELIGIBILITY:
Inclusion Criteria:

* Within the general population, all persons over 18 years of age living or working in the country Center Bretagne (including Pays Pays Ouest Bretagne, Pleyben and Callac) with a moderate cardiovascular risk score based on the Interheart clinical risk score (score 9-15).

Exclusion Criteria:

* Pregnancy
* Age under 18 years old
* Patient in secondary cardiovascular prevention
* Nobody living or working in Central Brittany (Pays Center Ouest Bretagne and Pays de Pleyben and Callac)
* Low (<9) or high cardiovascular risk score by Interheart score (> 15).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 583 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Measurement of the non laboratory Interheart risk score | 24 months
  Comparison of the Non Laboratory Interheart risk average score between the two arms at 24 months. This scale is used to predict incident cardiovascular disease.This score is summed and is calculated from questions about family history, type of diet and sports activities.

SECONDARY OUTCOMES:
Measurement of the quality of life | 24 months
  Quality of life evaluated by the World Health Organization Quality of Life (WHOQOL scale brief). This questionnaire contains two items from the Overall Quality of Life and General Health, and one item from each of the 24 facets included in The WHOQOL-100. It assesses the individual's perceptions in the context of their culture and value systems, and their personal goals, standards and concerns.The WHOQOL-BREF instrument comprises 26 items, which measure the following broad domains: physical health, psychological health, social relationships, and environment. The score is summed.
BMI | 24 months
  Reduction of BMI
Evaluation of the level of smoking | 24 months
  Reduction of the number of smokers / reduction of the number of cigarettes per smoker
Improvement of the diet | 24 months
  Improvement of the diet with the Dietary Approaches to Stop Hypertension Quality questionnaire (DASH-Q). This questionnaire was developed in 1997, emphasizing on 8 components: high consumption of fruits, vegetables, whole grains, low-fat dairy foods, legumes and nuts, and low intake of sodium, sweetened beverages, and red and processed meat. The total score is summed.
Level of physical activity | 24 months
  Level of physical activity by the International Physical Activity Questionnaire (IPAQ). This questionnaire comprises a set of 4 questionnaires. Long (5 activity domains asked independently) and short (4 generic items) versions for use by either telephone or self-administered methods are available. The purpose of the questionnaires is to provide common instruments that can be used to obtain internationally comparable data on health-related physical activity.The total score is summed.
Alcohol consumption | 24 months
  Alcohol consumption by collecting the reported weekly consumption of alcohol

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - LE GOFF, La Forest-Landerneau
  - LE RESTE, Lanmeur

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning five years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Derived] Le Goff D, Aerts N, Odorico M, Guillou-Landreat M, Perraud G, Bastiaens H, Musinguzi G, Le Reste JY, Barais M. Practical dietary interventions to prevent cardiovascular disease suitable for implementation in primary care: an ADAPTE-guided systematic review of international clinical guidelines. Int J Behav Nutr Phys Act. 2023 Jul 28;20(1):93. doi: 10.1186/s12966-023-01463-9. PMID 37507692
- [Derived] Le Goff D, Barais M, Perraud G, Derriennic J, Aujoulat P, Guillou-Landreat M, Le Reste JY. Innovative cardiovascular primary prevention population-based strategies: a 2-year hybrid type 1 implementation randomised control trial (RCT) which evaluates behavioural change conducted by community champions compared with brief advice only from the SPICES project (scaling-up packages of interventions for cardiovascular disease prevention in selected sites in Europe and sub-Saharan Africa). BMC Public Health. 2021 Jul 19;21(1):1422. doi: 10.1186/s12889-021-11443-y. PMID 34281516